CLINICAL TRIAL: NCT03424291
Title: A Retrospective Clinical Study of Apatinib in Combination With Radiotherapy / Chemotherapy Second-line and Above in the Treatment of Recurrent / Metastatic Head and Neck Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AHEAD-HNP016
Record Dates: First submitted 2018-01-31; First posted 2018-02-06 (Actual); Last update posted 2018-02-06 (Actual); Status verified 2017-07

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — apatinib; Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apatinib plus chemoradiation (Experimental): Apatinib 500 mg qd po Taxus + platinum or 5FU + platinum (drug dose reference to clinical) palliative radiotherapy dose ≥ 40Gy and radical radiotherapy dose (60-70Gy)
  Interventions: Drug: Apatinib plus chemoradiation

INTERVENTIONS:
Drug: Apatinib plus chemoradiation — Apatinib 500 mg qd po Taxus + platinum or 5FU + platinum (drug dose reference to clinical) palliative radiotherapy dose ≥ 40Gy and radical radiotherapy dose (60-70Gy)

SUMMARY:
The purpose of this study is to confirm the safety and efficacy of Apatinib in Combination With Radiotherapy / Chemotherapy for Second-line and Above Recurrent / Metastatic Head and Neck Squamous Cell Carcinoma.

DETAILED DESCRIPTION:
Head and neck cancer refers to the skull base to the supraclavicular, cervical spine within the scope of all malignant tumors is more common in China's malignant tumors. Head and neck cancer mainly surgery and radiotherapy, chemotherapy alone or in combination therapy, common head and neck squamous cell carcinoma chemotherapy programs are: PF regimen (cisplatin + 5-fluorouracil), PLF program (cisplatin + carboplatin +5 - fluorouracil), TPF program (cisplatin + 5 - fluorouracil + paclitaxel) and so on. The researcher consider to add apatinib,a tyrosine kinase inhibitor of VEGF,to the therapy of these patients.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 and ≤ 70 years of age.
2. Pathologically confirmed advanced head and neck squamous cell carcinoma, with measurable lesions (tumor lesions CT scan diameter ≥ 10mm, lymph node lesions CT scan short diameter ≥ 15mm, the scan layer thickness is not greater than 5mm, measurable after the lesion recurrence / metastasis Received radiotherapy, frozen and other local treatment).
3. Patients with recurrent or metastatic head and neck squamous cell carcinoma who have undergone radiotherapy and chemotherapy to treat disease progression.

   Note: adjuvant therapy within 6 months of recurrence, adjuvant therapy is defined as first-line treatment.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 2.
5. Life expectancy of more than 6 months.
6. Subjects underwent additional treatment of the damage recovered (NCI-CTCAE Version 4.0 Grading ≤ 1), where the interval between receiving nitrosourea or mitomycin was> 6 weeks; receiving other cytotoxic drugs, bevacizumab (Avastin), radiotherapy or surgery ≥ 4 weeks; EGFR TKI class of targeted drugs ≥ 2 weeks.
7. Adequate hepatic, renal, heart, and hematologic functions: ANC ≥ 1.5×109/L, PLT ≥ 80×109/L, HB ≥ 90 g/L, TBIL ≤ 1.5×ULN, ALT or AST

   ≤ 2.5×ULN (or ≤ 5×ULN in patients with liver metastases), Serum Cr ≤ 1.5×ULN, Cr clearance ≥ 45 mL/min.
8. Women of childbearing age must have had reliable contraception or have had a pregnancy test (serum or urine) within 7 days prior to enrollment with a negative result and would be prepared to use the appropriate method of contraception 8 weeks after the test and the last administration of the test drug. For males, consent is to be given to contraception or surgical sterilization 8 weeks after the test and the last administration of the test drug.
9. Signed the informed consent form prior to patient entry.

Exclusion Criteria:

1. Non-squamous cell carcinoma (including squamous cell carcinoma mixed with other pathological types), nasopharyngeal carcinoma.
2. Active brain metastases, meningococcal meningitis, patients with spinal cord compression, or imaging at CT or MRI examination revealed brain or pia mater disease（Patients who have completed treatment and whose symptoms are stable in the first 21 days of randomization may be enrolled in the study but may be diagnosed as having no intracerebral hemorrhage by MRI, CT or venography）.
3. Uncontrollable hypertension (systolic BP ≥140 mmHg or diastolic BP

   ≥90 mmHg, despite optimal medical therapy).
4. grade II The above myocardial ischemia or myocardial infarction, poor control of arrhythmia (including QTc interval male ≥ 450 ms, female ≥ 470 ms); NYHA standards, Ⅲ ~ Ⅳ grade cardiac insufficiency, or cardiac ultrasound examination prompted left ventricular ejection Score (LVEF) <50%.
5. Patients whose routine urine tests indicate that urine protein ≥ ++ or verifies that the 24-h urine protein quantitation ≥ 1.0 g.
6. Patients who had obvious hemoptysis within 2 months before screening, or experienced daily hemoptysis with a volume more than half a tea spoon (2.5ml) or above.
7. Coagulation dysfunction (INR> 1.5, PT> ULN +4s or APTT> 1.5 ULN), with bleeding tendency or ongoing thrombolysis or anti-blood coagulation treatment；Patients treated with anticoagulants or vitamin K antagonists such as warfarin, heparin, or the like.
8. Long-term, unhealed wounds or fractures.
9. Patients who have history of psychotropic substance abuse who can not be abstinent or who have mental disorders.
10. According to the researchers' judgment, there are other serious patients who are endangered or have concomitant diseases that affect the completion of the study.
11. Patients with CNS metastases.
12. Pregnant or lactating women.
13. Researchers think it is not suitable for inclusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-07-05 (Actual); Primary Completion 2018-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | up to 2 year
  From date of randomization until the date of first documented progression or date of death from any cause

SECONDARY OUTCOMES:
Overall survival(OS) | up to 2 year
  From date of randomization until the date of death from any cause
Objective Response Rate (ORR) | up to 1 year
  From date of randomization until the date of death from any cause
Disease Control Rate (DCR) | up to 1 year
  Defined as the proportion of patients with a documented complete response, partial response, and stable disease (CR
  + PR + SD)
Duration of response（DOR） | up to 2 year

CONTACTS AND LOCATIONS:
Overall Officials: hui Wu, Principal Investigator — Henan Cancer Hospital; wei Du, Principal Investigator — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China